CLINICAL TRIAL: NCT07258732
Title: Study on the Impact of Probiotics on Postoperative Gastrointestinal Symptoms and Gut Microbiota After Sleeve Gastrectomy: A Randomized-Control Trial
Brief Title: The Impact of Probiotics on Bariatric Treatment Outcomes
Acronym: PROBE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warmia and Mazury in Olsztyn (Other)
Responsible Party: Principal Investigator, Natalia Dowgiałło-Gornowicz, MD, PhD, Associate Professor, University of Warmia and Mazury in Olsztyn
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1/2024
Record Dates: First submitted 2025-07-10; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Obesity &Amp; Overweight
Keywords: obesity; sleeve gastrectomy; constipation
MeSH Terms: conditions — Obesity; Overweight; Constipation | interventions — Probiotics; Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Diet
- Control (Active Comparator)
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotics containing Bifidobacterium animalis AMT30, Bifidobacterium breve AMT32, and Lactobacillus plantarum AMT14.
  Arms: Control
Other: Diet — Placebo
  Arms: Placebo

SUMMARY:
The planned study aims to assess whether probiotics improve the quality of life in patients during the early postoperative period following sleeve gastrectomy, and whether they influence the absorption of micro- and macronutrients.

Patients eligible for inclusion will have a BMI of 40 kg/m² or higher and must have successfully completed the qualification process for sleeve gastrectomy. Exclusion criteria include chronic gastrointestinal diseases, antibiotic use within 4 weeks prior to surgery, and lack of consent to participate in the study.

On the day before surgery, a stool sample will be collected from each patient for microbiological analysis to assess the composition of gut bacteria. Patients will then undergo sleeve gastrectomy using a standard surgical technique.

After the operation, participants will be randomized into two groups. The first group will receive probiotics containing Bifidobacterium animalis AMT30, Bifidobacterium breve AMT32, and Lactobacillus plantarum AMT14. These strains are deposited in the Polish Collection of Microorganisms at the Polish Academy of Sciences in Wrocław and are protected by Polish, European, and U.S. patents. The second group will receive a placebo.

As part of follow-up, stool samples will be collected again one month and three months after surgery for comparative microbiological analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years.
2. BMI over 40 kg/m² or over 35 kg/m² with obesity-related comorbidities.
3. Successful qualification for sleeve gastrectomy.
4. Informed consent to participate in the study.

Exclusion Criteria:

1. Age under 18 years.
2. Chronic gastrointestinal diseases.
3. Use of antibiotic therapy within 4 weeks prior to surgery.
4. Lack of consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the impact of probiotics on the resolution of constipation after sleeve gastrectomy | one and three months after surgery
  The primary outcome of the study is to assess the effect of probiotics on the frequency of defecation in the early weeks following surgery. The patient would be asked whether constipation occurred (yes or no).

SECONDARY OUTCOMES:
Assessment of the impact of probiotics on gastrointestinal symptoms after SG | one and three months after surgery
  The secondary outcome of the study is to assess the effect of probiotics on the frequency of defecation in the early weeks following surgery. The patient would be asked about the number of stools passing per week.
Assessment of the impact of probiotics on gastrointestinal symptoms after SG | one and three months after surgery
  The secondary outcome of the study is to assess the effect of probiotics on the frequency of defecation in the early weeks following surgery. The patient would be asked about the subjective assessment of the ease of defecation.
  A Likert scale of 1-5 was used, where 1 indicated great difficulty with defecation, and 5 indicated no difficulty with defecation.
Assessment of the impact of probiotics on gastrointestinal symptoms after SG | one and three months after surgery
  The secondary outcome of the study is to assess the effect of probiotics on the frequency of defecation in the early weeks following surgery. The patient would be asked about the feeling of bowel movement completeness.
  A Likert scale of 1-5 was used, where 1 indicated a complete feeling of incomplete defecation, and 5 indicated a complete feeling of defecation.
Metabolic changes after the probiotics use in patients after SG | one and three months after surgery
  The secondary aim is to evaluate laboratory tests to identify any metabolic changes associated with probiotic use.
  It would be: Hemoglobin (Hb): g/dL
Metabolic changes after the probiotics use in patients after SG | one and three months after surgery
  The secondary aim is to evaluate laboratory tests to identify any metabolic changes associated with probiotic use.
  It would be: Creatinine: mg/dL
Metabolic changes after the probiotics use in patients after SG | one and three months after surgery
  The secondary aim is to evaluate laboratory tests to identify any metabolic changes associated with probiotic use.
  It would be: Total Protein: g/L
Metabolic changes after the probiotics use in patients after SG | one and three months after surgery
  The secondary aim is to evaluate laboratory tests to identify any metabolic changes associated with probiotic use.
  It would be: Total Cholesterol: mg/dL
Metabolic changes after the probiotics use in patients after SG | one and three months after surgery
  The secondary aim is to evaluate laboratory tests to identify any metabolic changes associated with probiotic use.
  It would be: HbA1c: %
Metabolic changes after the probiotics use in patients after SG | one and three months after surgery
  The secondary aim is to evaluate laboratory tests to identify any metabolic changes associated with probiotic use.
  It would be: Ferritin: µg/L (ng/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Warmia and Mazury, Olsztyn, Poland

IPD SHARING:
Plan to Share IPD: No